CLINICAL TRIAL: NCT05818072
Title: The Prevalence, Risk Factors and Optimal Biopsy Protocol of Barrett's Esophagus in Taiwan - A Prospective Randomized Study
Brief Title: The Prevalence, Risk Factors and Optimal Biopsy Protocol of BE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: E-DA Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EDAHS-111031
Record Dates: First submitted 2023-03-05; First posted 2023-04-18 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Barrett's Esophagus; Intestinal Metaplasia
Keywords: Barrett's Esophagus; Columnar-lined esophagus; Intestinal metaplasia
MeSH Terms: conditions — Barrett Esophagus | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One biopsy (Experimental): Obtain one biopsy specimen at the proximal part of the the longest columnar-lined esophagus for patients with suspected Barrett's Esophagus
  Interventions: Procedure: One biopsy; Device: Endoscopy
- Three biopsy (Active Comparator): Obtain three biopsy specimens at the proximal, middle and distal part of the longest columnar-lined esophagus for patients with suspected Barrett's Esophagus
  Interventions: Procedure: Three biopsy; Device: Endoscopy
- Seattle protocol (Sham Comparator): Obtain 4-quadrant biopsy specimens at intervals of every 1 to 2 cm throughout the the columnar-lined esophagus for patients with suspected Barrett's Esophagus
  Interventions: Procedure: Seattle protocol; Device: Endoscopy

INTERVENTIONS:
Procedure: One biopsy — To do one biopsy at the proximal part of the longest columnar-lined esophagus.
  Arms: One biopsy
Procedure: Three biopsy — To do three biopsy at the proximal, middle and distal part of the longest columnar-lined esophagus.
  Arms: Three biopsy
Procedure: Seattle protocol — To do 4-quadrant biopsy every 1-2 cm at the esophagogastric junction. Seattle protocol has been considered as the gold standard biopsy protocol for patients with suspected Barrett's Esophagus.
  Arms: Seattle protocol
Device: Endoscopy — The participants will receive meticulous endoscopic examination with narrow-band imaging.

SUMMARY:
Detections of goblet cells and dysplasia are crucial for diagnosis and determining the surveillance program of Barrett's esophagus (BE). However, the optimal biopsy numbers and their yield rates of intestinal metaplasia (IM) and dysplasia are still uncertain, especially in Asia. The aim of this study was to determine the optimal biopsy protocol of BE.

DETAILED DESCRIPTION:
Barrett's esophagus (BE) is premalignant lesion for esophageal adenocarcinoma (EAC) and defined as the distal esophageal squamous epithelium replaced by columnar epithelium with histologic confirmation of intestinal metaplasia (IM). The accurate prevalence of BE is difficult to assess because part of people with BE are asymptomatic. However, the prevalence of gastroesophageal reflux disease (GERD) which is the main factor associated with BE has increased almost 50% during the last 20 years. Meanwhile, the general population prevalence of BE is estimated to increase to 3-10% in Western countries. The systematic review and meta-analysis also reported an upward trend in prevalence of BE in Asian countries. BE is an important heathy issue to investigate in either Western or Asian countries.

The annual rate of developing esophageal adenocarcinoma is around 0.2% to 0.5% in patients with BE. However, the annual adenocarcinoma progression risk is different between the non-dysplastic Barrett's esophagus (NDBE), BE with low-grade dysplasia (LGD) and high-grade dysplasia (HGD). The annual incidence of esophageal adenocarcinoma is 0.33%, 0.54% and 6.58% in patients with NDBE, BE with LGD and HGD, respectively. Among patients with NDBE, patients with short segment BE (SSBE) have the lower rate of progression to EAC than those who with long segment BE (LSBE) (0.07% vs 0.25%). Therefore, endoscopic surveillance of patients with BE is recommended by clinical practice guideline.

Detections of goblet cells and dysplasia are crucial for diagnosis and determining the surveillance program of BE. According to the Seattle protocol which has been widely recommended by clinical practice guidelines, biopsy specimens should be obtained every one cm to two cm interval across the four quadrants of the columnar epithelium of esophagus. Fewer endoscopists adhered to this protocol in clinical practice because of its laboriousness and time consumption. Most of patients with BE were categorized as SSBE and SSBE seems to be more prevalent in Asian populations. As the report of previous study which reviewed the general prevalence of BE in Western and Asian general populations, the ratio of SSBE to LSBE was ranging from 1.8 to 17.4 in the Western countries and 1.7 to 103 in the Asian countries. It's more difficult to adhere to the protocol in patients with SSBE.

However, the optimal biopsy numbers and their yield rates of IM and dysplasia are still uncertain, especially in Asia. The investigators aimed to assess the biopsy numbers and yield rates of IM and dysplasia in patients with columnar-lined esophagus (CLE) to determine the optimal biopsy protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adults with columnar-lined esophagus

Exclusion Criteria:

* A prior history of endoscopic treatment for Barrett's Esophagus
* A prior history of upper gastrointestinal malignancy
* A prior history of total or subtotal gastrectomy
* Esophageal varices noted during the procedure
* Uncontrolled coagulopathy
* Taking antiplatelet drug or anticoagulant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The yield rate of intestinal metaplasia | Up to 7 days histologic confirmation
  Defined as the proportion of histologic confirmation of goblet cells

SECONDARY OUTCOMES:
The yield rate of dysplasia | Up to 7 days histologic confirmation
  Defined as the proportion of histologic confirmation of columnar-lined epithelium with dysplasia
Adverse events | From the date of procedure until any events, assessed up to 2 weeks
  Including bleeding and perforation
Procedure time | From forcep insertion to biopsy complete, assessed up to 1 minutes
  Defined as from forcep insertion to biopsy complete

CONTACTS AND LOCATIONS:
Locations (1):
- E-DA Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharma P. Barrett Esophagus: A Review. JAMA. 2022 Aug 16;328(7):663-671. doi: 10.1001/jama.2022.13298. PMID 35972481
- [Result] Richter JE, Rubenstein JH. Presentation and Epidemiology of Gastroesophageal Reflux Disease. Gastroenterology. 2018 Jan;154(2):267-276. doi: 10.1053/j.gastro.2017.07.045. Epub 2017 Aug 3. PMID 28780072
- [Result] Shiota S, Singh S, Anshasi A, El-Serag HB. Prevalence of Barrett's Esophagus in Asian Countries: A Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2015 Nov;13(11):1907-18. doi: 10.1016/j.cgh.2015.07.050. Epub 2015 Aug 7. PMID 26260107
- [Result] Desai TK, Krishnan K, Samala N, Singh J, Cluley J, Perla S, Howden CW. The incidence of oesophageal adenocarcinoma in non-dysplastic Barrett's oesophagus: a meta-analysis. Gut. 2012 Jul;61(7):970-6. doi: 10.1136/gutjnl-2011-300730. Epub 2011 Oct 13. PMID 21997553
- [Result] Singh S, Manickam P, Amin AV, Samala N, Schouten LJ, Iyer PG, Desai TK. Incidence of esophageal adenocarcinoma in Barrett's esophagus with low-grade dysplasia: a systematic review and meta-analysis. Gastrointest Endosc. 2014 Jun;79(6):897-909.e4; quiz 983.e1, 983.e3. doi: 10.1016/j.gie.2014.01.009. Epub 2014 Feb 17. PMID 24556051
- [Result] Rastogi A, Puli S, El-Serag HB, Bansal A, Wani S, Sharma P. Incidence of esophageal adenocarcinoma in patients with Barrett's esophagus and high-grade dysplasia: a meta-analysis. Gastrointest Endosc. 2008 Mar;67(3):394-8. doi: 10.1016/j.gie.2007.07.019. Epub 2007 Nov 28. PMID 18045592
- [Result] Hamade N, Vennelaganti S, Parasa S, Vennalaganti P, Gaddam S, Spaander MCW, van Olphen SH, Thota PN, Kennedy KF, Bruno MJ, Vargo JJ, Mathur S, Cash BD, Sampliner R, Gupta N, Falk GW, Bansal A, Young PE, Lieberman DA, Sharma P. Lower Annual Rate of Progression of Short-Segment vs Long-Segment Barrett's Esophagus to Esophageal Adenocarcinoma. Clin Gastroenterol Hepatol. 2019 Apr;17(5):864-868. doi: 10.1016/j.cgh.2018.07.008. Epub 2018 Aug 8. PMID 30012433
- [Result] Shaheen NJ, Falk GW, Iyer PG, Souza RF, Yadlapati RH, Sauer BG, Wani S. Diagnosis and Management of Barrett's Esophagus: An Updated ACG Guideline. Am J Gastroenterol. 2022 Apr 1;117(4):559-587. doi: 10.14309/ajg.0000000000001680. PMID 35354777
- [Result] Fitzgerald RC, di Pietro M, Ragunath K, Ang Y, Kang JY, Watson P, Trudgill N, Patel P, Kaye PV, Sanders S, O'Donovan M, Bird-Lieberman E, Bhandari P, Jankowski JA, Attwood S, Parsons SL, Loft D, Lagergren J, Moayyedi P, Lyratzopoulos G, de Caestecker J; British Society of Gastroenterology. British Society of Gastroenterology guidelines on the diagnosis and management of Barrett's oesophagus. Gut. 2014 Jan;63(1):7-42. doi: 10.1136/gutjnl-2013-305372. Epub 2013 Oct 28. PMID 24165758
- [Result] Abrams JA, Kapel RC, Lindberg GM, Saboorian MH, Genta RM, Neugut AI, Lightdale CJ. Adherence to biopsy guidelines for Barrett's esophagus surveillance in the community setting in the United States. Clin Gastroenterol Hepatol. 2009 Jul;7(7):736-42; quiz 710. doi: 10.1016/j.cgh.2008.12.027. Epub 2009 Jan 13. PMID 19268726
- [Result] Ronkainen J, Aro P, Storskrubb T, Johansson SE, Lind T, Bolling-Sternevald E, Vieth M, Stolte M, Talley NJ, Agreus L. Prevalence of Barrett's esophagus in the general population: an endoscopic study. Gastroenterology. 2005 Dec;129(6):1825-31. doi: 10.1053/j.gastro.2005.08.053. PMID 16344051
- [Result] Tseng PH, Lee YC, Chiu HM, Huang SP, Liao WC, Chen CC, Wang HP, Wu MS, Lin JT. Prevalence and clinical characteristics of Barrett's esophagus in a Chinese general population. J Clin Gastroenterol. 2008 Nov-Dec;42(10):1074-9. doi: 10.1097/MCG.0b013e31809e7126. PMID 18360296